CLINICAL TRIAL: NCT06635447
Title: A Phase IIIb Single Arm, 2 Cohorts Study Assessing the Efficacy and Safety of Capivasertib+ Fulvestrant as Treatment for Locally Advanced(Inoperable) or Metastatic Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) Breast Cancer Following Recurrence or Progression On or After Treatment With Endocrine Therapy in Chinese Patients
Brief Title: Capivasertib+Fulvestrant asTreatment for Locally Advanced(Inoperable) or Metastatic HR+/HER2- Breast Cancer in Chinese Patients
Acronym: CAPItrue
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3612R00016
Record Dates: First submitted 2024-09-09; First posted 2024-10-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HR+/HER2-ABC; disease recurrence/progression
MeSH Terms: conditions — Breast Neoplasms; Disease Progression | interventions — capivasertib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Capivasertib+Fulvestrant
  Interventions: Drug: Capivasertib; Drug: Fulvestrant
- Cohort 2 (Experimental): Capivasertib+Fulvestrant
  Interventions: Drug: Capivasertib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Capivasertib — 400 mg, oral, twice daily; 4 days on and 3 days off
  Other Names: AZD5363
Drug: Fulvestrant — Fulvestrant IV

SUMMARY:
This is a multi-center, two-cohorts, phase IIIb study of Capivasertib+Fulvestrant in HR+/HER2-ABC who had disease recurrence/progression following 1-2L endocrine therapy.

The Primary objective is to assess the efficacy of capi+ful by assessment of TFST (Time to first subsequent treatment) of PIK3CA/AKT1/PTEN-altered subgroup in cohort1.

DETAILED DESCRIPTION:
This study will enroll about 300 patients in 2 cohorts . Cohort1 will include patients without prior fulvestrant treated and Cohort2 will include patients who received fulvestrant as the first-line treatment and progression ≥6 months after the first dosing of fulvestrant. Approximately 195 patients will be enrolled in Cohort1 and 105 patients will be enrolled in Cohort2.

All patients will receive weekly capivasertib (400 mg, oral, twice daily; 4 days on and 3 days off) and fulvestrant (at the approved dose regimen [500 mg intramuscular injections on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter]). All patients will attend a screening visit a maximum of 28 days prior to the start of study treatment.

ELIGIBILITY:
Inclusion Criteria

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the clinical study protocol (CSP).
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
3. Patients must be aged ≥18 years at the time of signing the ICF
4. Adult females, pre- and/or post-menopausal, and adult males -Pre-menopausal (and peri-menopausal i.e., those that do not meet the criteria for post-menopausal defined below) women can be enrolled if amenable to treatment with an LHRH agonist. Patients are to have commenced concomitant treatment with LHRH agonist prior to or on Cycle 1, Day 1 and must be willing to continue on it for the duration of the study -Post-menopausal women are defined as: a)aged ≥60 years of age, or b)aged <60 years of age and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments/chemotherapy/ovarian suppression/tamoxifen or similar. These patients should also have serum oestradiol and follicle stimulating hormone (FSH) levels confirmed as being within the standard laboratory reference range for post-menopausal females, or c)documented bilateral oophorectomy
5. Histologically confirmed HR+/HER2- breast cancer determined from the most recent tumour sample (primary or metastatic), as per the American Society of Clinical Oncology and College of American Pathologists guideline recommendations. To fulfil the requirement of HR+ disease, a breast cancer must express ER with or without co-expression of progesterone receptor. 1)ER+ defined as ≥1% of tumour cells stain positive for ER on immunohistochemistry (IHC) or, if no percentage is available, then an Allred IHC score of ≥3/8, 2)Progesterone receptor positive defined as ≥1% of tumour cells stain positive for progesterone receptor on IHC or, if no percentage is available, then an Allred IHC score of ≥3/8; or progesterone receptor negative defined as <1% of tumour cells stain positive for progesterone receptor on IHC or, if no percentage is available, then an Allred IHC score of ≤2/8; or progesterone receptor unknown, 3)or the investigator assesses the condition as HR+ status and 4)HER2- defined as 0 or 1+ intensity on IHC, or 2+ intensity on IHC and no evidence of amplification on in situ hybridisation (ISH), or if IHC not done, no evidence of amplification on ISH.

   Metastatic or locally advanced disease with radiographic or objective evidence of recurrence or progression (cancer that has progressed during or after a recent treatment period).; locally advanced disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible) Patients are to have received treatment with an endocrine therapy containing regimen (single agent or in combination) and have: a)Radiological evidence of breast cancer recurrence or progression during treatment or within 12 months after the end of treatment with a neoadjuvant or adjuvant endocrine therapy, OR b)Radiological evidence of progression while on prior ET administered as a treatment line for locally advanced or metastatic breast cancer (this does not need to be the most recent therapy) (for patients with breast cancer recurrence or progression while on, or within 12 months of the end of (neo)adjuvant treatment with an ET will be limited to approximately 10%).
6. Patients must have at least 1 measurable lesion.
7. Patients must be eligible for fulvestrant therapy as per local investigator assessment.
8. Consent to submit and provide a mandatory FFPE tumour sample for central testing.
9. Patients must be able to swallow and retain oral medication.
10. Eastern Cooperative Oncology Group (ECOG)/ World Health Organisation (WHO) performance status 0 or 1 and life expectancy of ≥12 weeks.
11. Patients with PIK3CA/AKT1/PTEN alterations confirmed by central laboratory NGS testing. (Note: Applicable exclusively to patients enrolled under Protocol Version 2.0.)

Exclusion Criteria

1. A disease burden that makes the patient ineligible for endocrine therapy per the investigator's best judgement (e.g., symptomatic visceral disease that is potentially life-threatening in the short-term)
2. History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease. Radiotherapy within 2 weeks prior to the first dose of study intervention. Major surgery (excluding placement of vascular access) within 4 weeks prior to study treatment initiation
3. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment
4. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids within 4 weeks prior to study treatment initiation
5. Leptomeningeal metastase
6. Active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
7. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
8. Any of the following cardiac criteria: a)Mean resting QT interval corrected by Fridericia's formula (QTcF) >470 msec obtained from 3 consecutive ECGs b)History of QT prolongation associated with other medications that required discontinuation of that medication. - Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block) c)Medical history significant for arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted to enter the study based on the Investigator judgement with cardiologist consultation recommended. d)Any factors that increase the risk of corrected QT interval (QTc) prolongation or risk of arrhythmic events such as heart failure, clinically significant electrolyte abnormalities including hypokalaemia, hypomagnesaemia, and hypocalcaemia, potential for Torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval e)Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, myocardial infarction, unstable angina pectoris, f)Congestive heart failure New York Heart Association (NYHA) grade ≥2
9. Clinically significant abnormalities of glucose metabolism defined as HbA1c ≥8.0% (63.9 mmol/mol) at screening.

   Note: for any patient with evidence of impaired glucose control or insulin resistance refer to the Capivasertib Toxicity Management Guidelines.
10. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: a)Absolute neutrophil count <1.5 × 109/L b)Platelet count <100 × 109/L c)Haemoglobin <9 g/dL (<5.59 mmol/L). [NOTE: any blood transfusion must be >14 days prior to the determination of a haemoglobin ≥9 g/dL (≥5.59 mmol/L)] d)Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) >2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or >5 × ULN in the presence of liver metastases e)Total bilirubin >1.5 × ULN (Patients with confirmed Gilbert's syndrome may be included in the study) f)Creatinine >1.5 × ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault formula (using actual body weight) without the need for chronic dialysis therapy.
11. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, or active infection
12. Known HIV infection that is not well controlled. (All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load, CD4+ count of >350, no history of AIDS-defining opportunistic infection within the past 12 months, and on anti-HIV medications for at least 4 weeks. Teams should consider adding appropriate information into sections for AE monitoring and the concomitant medication tables.[HIV inclusion criteria may be adjusted to lower CD4+ count values if clinically indicated if the patient has a potentially curable malignancy or for interventions in a later stage of development that have demonstrated prior activity within a given cancer, please adjust if necessary.])
13. Known active hepatitis B or C infection, positive hepatitis C antibody, positive hepatitis B virus surface antigen. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients receiving antiretroviral therapies which are strong inhibitors or inducers of CYP3A4 will be excluded due to the potential for drug-drug interaction with capivasertib as per Table 19 Drug Interactions that affect Capivasertib.
14. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of fulvestrant or LHRH agonist (if applicable)
15. Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib
16. Previous allogenic bone marrow or solid organ transplant
17. Known immunodeficiency syndrome
18. History of hypersensitivity to active or inactive excipients of capivasertib, fulvestrant and LHRH agonists (if applicable, i.e., concomitant LHRH agonist required in this study) or drugs with a similar chemical structure or class to capivasertib, fulvestrant or LHRH agonists (if applicable, i.e., concomitant LHRH agonist required in this study)
19. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
20. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
21. More than 2 lines of endocrine therapy for inoperable locally advanced or metastatic disease in Cohort 1; More than 1 lines endocrine therapy for inoperable locally advanced or metastatic disease in Cohort2 For Cohort 2, Patients must receive fulvestrant ≤ 1L endocrine treatment for ABC and progression <6 months after the first dosing of fulvestrant.

    For patients with breast cancer recurrence or progression while on, or within 12 months of the end of (neo)adjuvant treatment with an ET will be limited to approximately 10%.

    NOTE: If an attempt to downstage a locally advanced tumour with endocrine therapy was made in the absence of metastatic breast cancer (neoadjuvant), and the tumour operated upon, then this does not count as a line of therapy for ABC. In contrast, if the tumour remained inoperable, this treatment should be included as a line of therapy for ABC. Adjuvant endocrine therapy is not considered a line of therapy for ABC. In addition, switching drugs within a line of therapy to manage toxicities in the absence of progressive disease does NOT count as a new line of therapy.
22. More than 1 line of chemotherapy for inoperable locally advanced or metastatic disease (Patients experienced recurrence or progression during chemotherapy of ABC will be limited to a maximum approximately of 15% of the total study population; once this limit is met the enrolment of this group of patients should be terminated). Adjuvant and neoadjuvant chemotherapy are not classed as lines of chemotherapy for ABC
23. Prior treatment with any of the following: a)AKT, PI3K and mTOR inhibitors b)Fulvestrant, and other SERDs in Cohort1 c)Nitrosourea or mitomycin C within 6 weeks prior to study treatment initiation d)Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents within 3 weeks prior to study treatment initiation. A longer washout period may be required for drugs with a long half-life (e.g., biologics) as agreed by the sponsor e)Systemic therapy: Prior exposure to any chemotherapy or anti-cancer agents other than those specified in the protocol (e.g. hormonal therapy such as LHRH agonists) without appropriate washout period before enrolment, for example, enrolment within 3 half-lives of a small molecule anti-cancer agent, or within 4 weeks for any antibody-based anticancer agents. f)Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort) or drugs that are sensitive to CYP3A4 inhibition within 1 week prior to study treatment initiation. g)Any concomitant medication that may interfere with fulvestrant safety and efficacy based on the prescribing information of fulvestrant and local clinical guidelines.
24. Participation in another clinical study with a non-marketed investigational medicinal product (IMP) administered in the last 30 days or 5 half-lives, whichever is longer (for IMPs which are a previously marketed drug, regardless of indication.)
25. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
26. Pregnant women (confirmed with positive pregnancy test) or breast-feeding women or women who are planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Time to first subsequent treatment (TFST) of PIK3CA/AKT1/PTEN-altered population in Cohort 1 | From the first dose of study intervention to the earlier of start date of the first subsequent therapy after discontinuation of study intervention, or death in PIK3CA/AKT1/PTEN-altered population in Cohort 1, up to approximately 2 years
  To assess the efficacy of capi+ful by assessment of TFST (Time to first subsequent treatment) of PIK3CA/AKT1/PTEN-altered subgroup in cohort1

SECONDARY OUTCOMES:
Progression-free survival (PFS) in PIK3CA/AKT1/PTEN-altered population in Cohort 1 and 2 | From the first dose until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from study treatment or receives another anti-cancer therapy prior to progression
  To assess the efficacy of capi+ful by assessment of PFS of PIK3CA/AKT1/PTEN-altered population in Cohort 1 and 2
Time to first subsequent treatment (TFST) in PIK3CA/AKT1/PTEN-altered population in Cohort 2 | From the first dose of study intervention to the earlier of start date of the first subsequent therapy after discontinuation of study intervention, or death in PIK3CA/AKT1/PTEN-altered population in Cohort 2, up to approximately 2 years
  To assess the efficacy of capi+ful by assessment of TFST in PIK3CA/AKT1/PTEN-altered population in Cohort 2
Number of participants with AEs/SAEs | From time of signature of the ICF, throughout the treatment period and including the 30-day follow-upperiod after discontinuation of study drug, up to approximately 2 years
  To assess the safety and tolerability of capivasertib + fulvestrant in cohort1 and cohort2
Objective response rate (ORR) in PIK3CA/AKT1/PTEN-altered population in Cohort 1 and 2 | The percentage of PIK3CA/AKT1/PTEN-altered subjects with at least one investigator-assessed response of CR or PR and will be based on a subset of all PIK3CA/AKT1/PTEN-altered subjects with measurable disease at baseline per the site investigator.
  To assess the efficacy of capi+ful by assessment of ORR of PIK3CA/AKT1/PTEN-altered population in Cohort 1 and 2
Number of participants with AEs/SAEs in PIK3CA/AKT1/PTEN-altered population | From time of signature of the ICF, throughout the treatment period and including the 30-day follow-upperiod after discontinuation of study drug in PIK3CA/AKT1/PTEN-altered population, up to approximately 2 years
  To assess the safety and tolerability of capivasertib + fulvestrant of PIK3CA/AKT1/PTEN-altered population in Cohort 1 and Cohort 2

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, PhD, Principal Investigator — Clinical Trial Ethics Committee of The Fifth Medical Center of the Chinese People's Liberation Army General Hospital
Locations (54):
- China (54):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Deyang
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Jining
  - Research Site, Kashgar
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Meizhou
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Sichuan
  - Research Site, Suining Shi
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tangshan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wanzhou
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient- level data from AstraZeneca group of companies sponsored clinical trials via the request portal. Plan Description: All request will be evaluated as per the Az disclosure commitment: https://astrazenecaarouptrials.pharmacm.com/ST/Submission/Disclosure Yes. indicates that Az are accepting requests for IPD ,but this does not mean are quests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment at made to the EFPIA Pharma Data Sharing Principles .For details of our timeline please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement(non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to a air access. For additional details. please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home